CLINICAL TRIAL: NCT06568211
Title: VRx@Home: A Virtual Reality At-Home Intervention for Persons Living With Dementia and Their Care Partners
Brief Title: A Virtual Reality at Home Intervention for People Living With Dementia
Acronym: VRx@Home
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AGE-WELL, Inc (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Associated Medical Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-5701; 163902 (Other Grant/Funding Number: Canadian Consortium on Neurodegeneration in Aging Grant)
Record Dates: First submitted 2024-08-14; First posted 2024-08-23 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-08

CONDITIONS: Dementia
Keywords: Virtual Reality; Tablet; Reminiscence; Verbal communication; Nonverbal communication; Interpersonal Relationship; Quality of Life; Well-Being; Person Living with Dementia; Care Partner
MeSH Terms: conditions — Dementia; Nonverbal Communication | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: VR first (Experimental): Those assigned to Group A will be placed in the Virtual Reality (VR) intervention phase first. All participants will begin with a baseline picture book condition (week 0), and then those in Group A, will complete the VR intervention condition in the first two weeks (weeks 1 & 2). After completing the two weeks of VR intervention, participating families will be asked to complete a set of standardized questionnaires. The following next two weeks (weeks 3 & 4), participants will complete the Tablet-only intervention phase. At the end of this phase, participating families will again complete the same standardized questionnaires and will participate in a semi-structured interview about their experiences. Each session is expected to include 20 minutes of VR exposure. Each session will also be video-recorded for later analyses.
  Interventions: Device: Virtual Reality; Device: Tablet-Only
- Group B: Tablet-only first (Experimental): Those assigned to Group B will be placed in the Tablet-only intervention phase first. All participants will begin with a baseline picture book condition (week 0), and then those in Group B, will complete the Tablet-only condition in the first two weeks (weeks 1 & 2). After completing the two weeks of Tablet-only intervention, participating families will be asked to complete a set of standardized questionnaires. The following next two weeks (weeks 3 & 4), participants will complete the VR intervention phase. At the end of this phase, participating families will again complete the same standardized questionnaires and will participate in a semi-structured interview about their experiences. Each session is expected to include 20 minutes of VR exposure. Each session will also be video-recorded for later analyses.
  Interventions: Device: Virtual Reality; Device: Tablet-Only

INTERVENTIONS:
Device: Virtual Reality — Persons living with dementia (PLwD) will view 360-degree videos using a commercially-available Virtual Reality (VR) head mounted display that has built-in speakers. While wearing the VR headset, PLwD-participant will be able to visually explore the virtual environments by turning their head to face different directions. Care partner-participants will take part in the VR experience concurrently by viewing a tablet that is connected to the VR headset through the "screen mirroring" function.
  Other Names: VR; HMD
Device: Tablet-Only — PLwD and care partner will view 360-degree videos together on a commercially-available tablet that has built-in speakers. They will be able to visually explore the virtual environment using the touch screen (dragging the view around with their fingers).
  Other Names: Tablet

SUMMARY:
The goal of the current study is to design and evaluate a virtual reality (VR) at-home intervention to facilitate communication between persons living with dementia (PLwD) and their family/friend care partners, and in turn improve their interpersonal relationships and quality of life. The project also aims to provide a direct comparison of an immersive VR system with non-immersive tablet-based technology.

PLwD and care partner interactions will be recorded during each of the following sessions and then used for the primary measure of verbal and non-verbal communication.

* Picture Book condition (baseline): PLwD and care partner view pictures together on photo album
* VR condition: PLwD watch 360 degree videos on a VR and the care partner watches the same content concurrently on a paired tablet
* Table-Only condition: PLwD and care partner watch 360 videos together on the tablet

DETAILED DESCRIPTION:
Head Mounted VR headsets allow a person to transport to alternate realities such as visiting another country, attending a concert or a sporting event. The evidence to date suggests that VR experiences have positive impact on the well-being of individuals living with dementia. Most of this work however, has been in more formal settings whether it's long-term care or community programs, with trained formal care partners or researchers. Further, little work has explored specifically communication outcomes within the family dynamics.

After obtaining informed consent, participants will complete a Demographic and Health History questionnaire, and then will be scheduled for their first home visit. During this session, researcher will provide training on how to use the devices, how to video-record the study sessions, and how to complete study questionnaires through the supplied laptop. The PLwD and care partner will also view a picture book together while their interaction is being recorded through a video-conferencing software.

Participants will then begin the four weeks of intervention, where they will either be placed in the VR first intervention condition for the first two week or the Tablet-only first intervention condition (weeks 1 and 2), and then they will switch and receive the other device in the following two weeks (weeks 3 and 4). Participants will receive additional at-home training in-between two intervention phases. Irrespective of the condition, once a week participants will have a session with researcher over a video-conferencing software, where they watch a 20 mins video sequence that has a combination of 4 videos of different themes (animal, entertainment, travel, and sports) preselected for them. This is then followed by a short semi-structured interview asking participants about their preferences and experience. In addition, participants are asked to try the devices on their own and record their interactions.

In addition to the video recording of sessions which will be used for analyses of verbal and non-verbal communication, and interview data, participants will be asked to complete a set of questionnaires at baseline, and after each phase of the intervention. They will also be given a journal to note down any additional information they would like to share beyond those captures in interviews and questionnaires.

After completing the study, a final semi-structure interview will be conducted with participants to evaluate the overall feasibility and effectiveness of intervention. Study will complete with a final home visit to pick up devices.

ELIGIBILITY:
Given the nature of the study, the participating dyads will be required to have access to high-speed internet with a reliable WiFi connection. Additional inclusion/exclusion criteria are as follows:

PLwD inclusion criteria:

* report having dementia
* currently living at home

PLwD exclusion criteria:

* recent history of seizure, epilepsy, head trauma, or stroke
* pacemaker
* cervical conditions or injuries
* open face wounds
* alcohol-related dementia/Korsakoff syndrome
* having a Public Guardian and Trustee as substitute decision maker

Care partner inclusion criteria:

* identify as one of the primary care partners for the PLwD
* able to speak and understands English
* 18 years and older

Care partner exclusion criteria:

* professional/formal care partners for the PLwD
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Quality of conversation and dyadic interactions (observations) | Measures will be collected from baseline until the end of the intervention (week 4).
  Trained research assistants will code the video recordings for the quality of participation, support, and engagement using the standardized Measure of Participation in Conversation for Dementia (focused on PLwD) and Measure of Support in Conversation for Dementia (focused on Care partner).
Quality of conversation and dyadic interactions (self-report) | Measures will be collected from baseline until the end of the intervention (week 4).
  Participating families will complete a communication questionnaire.
Verbal Communication | Measures will be collected from baseline through the end of intervention (week 4)
  Trained research assistants will code the video recordings for measures of verbal communication (e.g., utterance length, coherence, reminiscence). This data will be analyzed through both qualitative and quantitative methods.
Nonverbal Communication | Measures will be collected from baseline through the end of intervention (week 4)
  Trained research assistants will code the video recordings for measures of nonverbal communication (e.g., gestures, familial expressions). This data will be analyzed through both qualitative and quantitative methods.

SECONDARY OUTCOMES:
Quality of Life | Measured at baseline, and after each phase of the intervention (end of week 2, and week 4)
  The Quality of Life in Alzheimer's Dementia (QoL-AD) will be administered to participants with dementia and caregiver-participants to evaluate subjective quality of life. The QoL-AD is a 13-item questionnaire employing 4-point Likert scales. Higher scores indicate greater subjective quality of life.
Well-Being | Measured at baseline, and after each phase of the intervention (end of week 2, and week 4)
  The WHO (Five) Well-Being Index will be administered to participants living with dementia and caregiver-participants to evaluate subjective wellbeing. The WHO (Five) is a 5-item questionnaire employing 6-point Likert scales.
Caregiver Burden | Measured at baseline, and after each phase of the intervention (end of week 2, and week 4)
  The Short Zarit Burden Interview tool will be completed by caregiver-participants and will be used to evaluate subjective feelings of caregiver burden associated with being a caregiver for the person with dementia. The Short Zarit Burden Interview is a 6-item questionnaire that employs a 5-point Likert scale.
Usability/Preference | Measure will be collected after each phase of the intervention (end of week 2 and week 4)
  System Usability Scale (SUS) will be administered to evaluate device usability/ease-of-use for both VR and Tablet-only conditions. The SUS is a 10-item questionnaire employing 5-point Likert scales.

CONTACTS AND LOCATIONS:
Locations (1):
- KITE Research Institute, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang LC, Yang YH. The Long-term Effects of Immersive Virtual Reality Reminiscence in People With Dementia: Longitudinal Observational Study. JMIR Serious Games. 2022 Jul 25;10(3):e36720. doi: 10.2196/36720. PMID 35877169
- [Background] Coelho T, Marques C, Moreira D, Soares M, Portugal P, Marques A, Ferreira AR, Martins S, Fernandes L. Promoting Reminiscences with Virtual Reality Headsets: A Pilot Study with People with Dementia. Int J Environ Res Public Health. 2020 Dec 12;17(24):9301. doi: 10.3390/ijerph17249301. PMID 33322679
- [Background] Appel L, Ali S, Narag T, Mozeson K, Pasat Z, Orchanian-Cheff A, Campos JL. Virtual reality to promote wellbeing in persons with dementia: A scoping review. J Rehabil Assist Technol Eng. 2021 Dec 21;8:20556683211053952. doi: 10.1177/20556683211053952. eCollection 2021 Jan-Dec. PMID 35024166
- [Background] Appel L, Appel E, Kisonas E, Lewis-Fung S, Pardini S, Rosenberg J, Appel J, Smith C. Evaluating the Impact of Virtual Reality on the Behavioral and Psychological Symptoms of Dementia and Quality of Life of Inpatients With Dementia in Acute Care: Randomized Controlled Trial (VRCT). J Med Internet Res. 2024 Jan 30;26:e51758. doi: 10.2196/51758. PMID 38289666
- [Background] Appel L, Appel E, Bogler O, Wiseman M, Cohen L, Ein N, Abrams HB, Campos JL. Older Adults With Cognitive and/or Physical Impairments Can Benefit From Immersive Virtual Reality Experiences: A Feasibility Study. Front Med (Lausanne). 2020 Jan 15;6:329. doi: 10.3389/fmed.2019.00329. eCollection 2019. PMID 32010701
- [Derived] Saryazdi R, Appel L, Lewis-Fung S, Carsault LA, Qi D, Garcia-Giler E, Campos JL. VRx@Home protocol: A virtual reality at-home intervention for persons living with dementia and their care partners. BMJ Open. 2024 Dec 20;14(12):e085442. doi: 10.1136/bmjopen-2024-085442. PMID 39806619